CLINICAL TRIAL: NCT05471596
Title: Prospective Analysis of In Vivo Laparoscopic Microwave Ablation Thermodynamics in Hepato-Pancreato-Biliary Solid Tumors
Brief Title: Prospective Analysis of In Vivo Laparoscopic Microwave Ablation Thermodynamics
Acronym: MWA
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00082683; 02-22-19E (Other: Atrium)
Record Dates: First submitted 2022-07-20; First posted 2022-07-25 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Liver Diseases
Keywords: Liver Cancer; Liver Lesion; Microwave Ablation; NeuWave Surgical; Hepatobiliarypancreato Surgery; Hepato-Pancreato-Biliary (HPB) Surgery
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- NeuWave Microwave Ablation System: Patients who underwent a Microwave Ablation at a participating institution and a NeuWave generator was utilized.
  Interventions: Device: NeuWave Microwave Ablation System

INTERVENTIONS:
Device: NeuWave Microwave Ablation System — The NEUWAVE System supports target ablation or linear coagulation in surgical liver resection procedures. The System offers a versatile probe portfolio, multi-probe synchrony and CO2 cooling to help control the shape, size and burn pattern of your ablations.

SUMMARY:
To prospectively collect and evaluate pre-operative, intra-operative, and post-operative variables for all patients undergoing surgical microwave ablation. All patients who have a surgical microwave ablation with the Neuwave system will be added to the database after their treatment and procedures have been completed.

DETAILED DESCRIPTION:
To prospectively collect and evaluate pre-operative, intra-operative, and post-operative variables for all patients undergoing surgical microwave ablation. All patients who have a surgical microwave ablation with the Neuwave system will be added to the database after their treatment and procedures have been completed. All data points will be collected from the electronic medical records (EMR) (office visit notes, operative notes, follow-up visits, CT scans, etc.). The collected data points will be utilized to study outcomes such as local/regional reoccurrences and distant occurrences related to hepatic tumor(s), whether there was complete destruction, residual disease/incomplete destruction, or recurrence at the ablation site. Overall-complications, length of stay, readmission rates, and any additional outcomes data that is relevant to MWA and improving surgical outcomes will also be collected.

There are various Microwave Ablation (MWA) systems available that are utilized at the study locations to treat hepatic tumors. For this study, the focus is on subjects treated with the Certus 140TM system from NeuWave Medical®. Certus 140TM microwave generator possesses a 2.45 gigahertz (GHz) operating frequency and can power up to 140 watts. It can deliver microwave energy through three distinct channels simultaneously through a single system and uses three distinct antenna types (LK, SR, PR). It also contains a CO2-based cooling system that helps limit the temperature of the handle and cable. It is compatible with a variety of probes (LK, SR and PR antenna) and offers two modes, Ablation mode and Surgical mode. The Ablation mode is used for ablating a substantial target for several minutes until the object of the ablation is necrotic. Surgical Mode is used to ablate or coagulate a target for shorter periods of time while frequently moving the probe in a technique known as "planar coagulation."

Current data and manufacturer guidelines for recommended ablation energy outputs for microwave ablation systems are obtained via ex vivo and animal models with tissues that exhibit different properties of energy transference than in vivo human tissues, particularly, human hepatic solid tumors. The objective is to prospectively assess the thermodynamics of microwave ablation energy in this context, specifically through the creation of power/time curves to predict future ablation volumes through single applications of MWA energy per lesion.

ELIGIBILITY:
Inclusion Criteria:

* Adults with hepatic tumors (Age >18 years or older)
* Treatment included microwave ablation with the Neuwave system

Exclusion Criteria:

* Age <18
* Benign Tumors
* Patients whose initial treatment plan did not include MWA, although they later received one (rescue MWA)
* Multiple tumors with distances or geometric relations rendering volumetrics incalculable or unduly confounded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (Age >18 years old) with hepatic lesion(s) treated by microwave ablation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Prospective Power/Time Analysis of In Vivo Laparoscopic Microwave Ablation Thermodynamics in Hepato-Pancreato-Biliary Sold Tumors Utilizing a Single Generator at a Single Surgical Center | Year 2
  The primary objective is to prospectively assess the thermodynamics of microwave ablation energy in this context, specifically through the creation of power/time curves to predict future ablation volumes through single applications of MWA energy per lesion.

SECONDARY OUTCOMES:
Liver appearance | Baseline
  Investigator to describe the appearance of the liver intraoperatively
Presence of extrahepatic disease | Baseline
  Investigator to describe if any extrahepatic disease is present
Chronic Liver Disease Evidence | Baseline
  Investigator to describe if any chronic liver disease is present
Number of Lesions | Baseline
  Number of lesions present
Lesion location | Baseline
  Location (segment) of each lesion
Size of Lesion | Baseline
  Size of each lesion
Amount of Power used | Baseline
  Power (W) used to ablate each lesion
Amount of Time used | Baseline
  Time (min) used to ablate each lesion
Distance between lesions | Baseline
  The distance between liver lesions
Ablation Dimensions | day 90
  Ablation dimensions as assessed by post-operative cross-sectional imaging using the x-axis along the length of the antenna tract and y-axis perpendicular to the antenna tract
Disease Recurrence Rate | week 4
  Disease recurrence defined as the radiologic presence of disease present at the index location at the 4-week follow up postoperative cross-sectional imaging
Number of New lesions | day 90
  New lesions noted on CT (as above) and their measurements
Radiographic liver appearance | day 90
  Liver appearance on CT
Radiographic extrahepatic disease | day 90
  Presence of extrahepatic disease on CT
Tumor measurement | Baseline
  Index tumor diameter and volume
Ablation Time | Baseline
  The time at which ablation occurred
Ablation Energy output | Baseline
  Energy output from ablation
Ablation Margins | day 90
  Ablation margins
Operative Time Amount | Baseline
  Time from first incision until final skin closure
Length of Stay | up to 90 days
  Time from hospital admission until hospital discharge
Readmission Rates | day 90
  Percentage of patients who were readmitted to the hospital after MWA
30 day complication rate | day 30
  Percentage of patients who experienced a complication 30 following MWA
90 day complication rate | day 90
  Percentage of patients who experienced a complication 90 following MWA

CONTACTS AND LOCATIONS:
Overall Officials: David A Iannitti, MD, Principal Investigator — Physician
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathur AK, Ghaferi AA, Sell K, Sonnenday CJ, Englesbe MJ, Welling TH. Influence of body mass index on complications and oncologic outcomes following hepatectomy for malignancy. J Gastrointest Surg. 2010 May;14(5):849-57. doi: 10.1007/s11605-010-1163-5. Epub 2010 Feb 6. PMID 20140536
- [Background] Groeschl RT, Pilgrim CH, Hanna EM, Simo KA, Swan RZ, Sindram D, Martinie JB, Iannitti DA, Bloomston M, Schmidt C, Khabiri H, Shirley LA, Martin RC, Tsai S, Turaga KK, Christians KK, Rilling WS, Gamblin TC. Microwave ablation for hepatic malignancies: a multiinstitutional analysis. Ann Surg. 2014 Jun;259(6):1195-200. doi: 10.1097/SLA.0000000000000234. PMID 24096760
- [Background] Swan RZ, Sindram D, Martinie JB, Iannitti DA. Operative microwave ablation for hepatocellular carcinoma: complications, recurrence, and long-term outcomes. J Gastrointest Surg. 2013 Apr;17(4):719-29. doi: 10.1007/s11605-013-2164-y. Epub 2013 Feb 13. PMID 23404173
- [Background] Bhardwaj N, Strickland AD, Ahmad F, El-Abassy M, Morgan B, Robertson GS, Lloyd DM. Microwave ablation for unresectable hepatic tumours: clinical results using a novel microwave probe and generator. Eur J Surg Oncol. 2010 Mar;36(3):264-8. doi: 10.1016/j.ejso.2009.10.006. Epub 2009 Oct 31. PMID 19880269
- [Background] Iannitti DA, Martin RC, Simon CJ, Hope WW, Newcomb WL, McMasters KM, Dupuy D. Hepatic tumor ablation with clustered microwave antennae: the US Phase II trial. HPB (Oxford). 2007;9(2):120-4. doi: 10.1080/13651820701222677. PMID 18333126
- [Background] Martin RC, Scoggins CR, McMasters KM. Safety and efficacy of microwave ablation of hepatic tumors: a prospective review of a 5-year experience. Ann Surg Oncol. 2010 Jan;17(1):171-8. doi: 10.1245/s10434-009-0686-z. Epub 2009 Aug 26. PMID 19707829
- [Background] Liang P, Wang Y, Yu X, Dong B. Malignant liver tumors: treatment with percutaneous microwave ablation--complications among cohort of 1136 patients. Radiology. 2009 Jun;251(3):933-40. doi: 10.1148/radiol.2513081740. Epub 2009 Mar 20. PMID 19304921
- [Background] Livraghi T, Meloni F, Solbiati L, Zanus G; Collaborative Italian Group using AMICA system. Complications of microwave ablation for liver tumors: results of a multicenter study. Cardiovasc Intervent Radiol. 2012 Aug;35(4):868-74. doi: 10.1007/s00270-011-0241-8. Epub 2011 Aug 11. PMID 21833809
- [Background] Laeseke PF, Lee FT Jr, van der Weide DW, Brace CL. Multiple-Antenna Microwave Ablation: Spatially Distributing Power Improves Thermal Profiles and Reduces Invasiveness. J Interv Oncol. 2009;2(2):65-72. PMID 21857888
- [Background] Harari CM, Magagna M, Bedoya M, Lee FT Jr, Lubner MG, Hinshaw JL, Ziemlewicz T, Brace CL. Microwave Ablation: Comparison of Simultaneous and Sequential Activation of Multiple Antennas in Liver Model Systems. Radiology. 2016 Jan;278(1):95-103. doi: 10.1148/radiol.2015142151. Epub 2015 Jul 2. PMID 26133361
- [Background] Knavel EM, Hinshaw JL, Lubner MG, Andreano A, Warner TF, Lee FT Jr, Brace CL. High-powered gas-cooled microwave ablation: shaft cooling creates an effective stick function without altering the ablation zone. AJR Am J Roentgenol. 2012 Mar;198(3):W260-5. doi: 10.2214/AJR.11.6503. PMID 22358023
- [Background] Poulou LS, Botsa E, Thanou I, Ziakas PD, Thanos L. Percutaneous microwave ablation vs radiofrequency ablation in the treatment of hepatocellular carcinoma. World J Hepatol. 2015 May 18;7(8):1054-63. doi: 10.4254/wjh.v7.i8.1054. PMID 26052394
- [Background] Al-Hakim RA, Abtin FG, Genshaft SJ, Kutay E, Suh RD. Defining New Metrics in Microwave Ablation of Pulmonary Tumors: Ablation Work and Ablation Resistance Score. J Vasc Interv Radiol. 2016 Sep;27(9):1380-1386. doi: 10.1016/j.jvir.2016.05.026. PMID 27566426
- [Background] Deshazer G, Merck D, Hagmann M, Dupuy DE, Prakash P. Physical modeling of microwave ablation zone clinical margin variance. Med Phys. 2016 Apr;43(4):1764. doi: 10.1118/1.4942980. PMID 27036574
- [Background] Liu D, Brace CL. Numerical simulation of microwave ablation incorporating tissue contraction based on thermal dose. Phys Med Biol. 2017 Mar 21;62(6):2070-2086. doi: 10.1088/1361-6560/aa5de4. Epub 2017 Feb 2. PMID 28151729
- [Background] Hubner F, Schreiner R, Reimann C, Bazrafshan B, Kaltenbach B, Schussler M, Jakoby R, Vogl TJ. Ex vivo validation of microwave thermal ablation simulation using different flow coefficients in the porcine liver. Med Eng Phys. 2019 Apr;66:56-64. doi: 10.1016/j.medengphy.2019.02.007. Epub 2019 Feb 28. PMID 30826254
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912